CLINICAL TRIAL: NCT02081326
Title: Repeat BCG Vaccinations for the Treatment of Established Type 1 Diabetes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Denise Louise Faustman, MD, Denise Louise Faustman, MD, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P002633
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type One; Diabetes Mellitus, Type I; Autoimmune Diabetes; Covid19
Keywords: Diabetes Mellitus, Type One; Diabetes Mellitus, Type I; Autoimmune Diabetes; Insulin Dependent Diabetes Mellitus 1; IDDM; COVID-19
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bacillus Calmette-Guérin (Experimental): 2 BCG vaccinations spaced 4 weeks apart during the first year and then 1 vaccination every year for the next 4 years
  Interventions: Biological: Bacillus Calmette-Guérin
- Saline injection (Placebo Comparator): 2 injections spaced 4 weeks apart during the first year, then 1 injection per year for the next 4 years
  Interventions: Biological: Saline injection

INTERVENTIONS:
Biological: Bacillus Calmette-Guérin — 2 BCG vaccinations spaced 4 weeks apart during the first year and then 1 vaccination every year for the next 4 years
  Arms: Bacillus Calmette-Guérin
Biological: Saline injection — 2 injections spaced 4 weeks apart during the first year, then 1 injection per year for the next 4 years
  Arms: Saline injection

SUMMARY:
The purpose of this study is to see if repeat bacillus Calmette-Guérin (BCG) vaccinations can confer a beneficial immune and metabolic effect on Type 1 diabetes. Published Phase I data on repeat BCG vaccinations in long term diabetics showed specific death of some of the disease causing bad white blood cells and also showed a short and small pancreas effect of restored insulin secretion. In this Phase II study, the investigators will attempt to vaccinate more frequently to see if these desirable effects can be more sustained.

Eligible volunteers will either be vaccinated with BCG in a repeat fashion over a period of four years, or receive a placebo treatment. The investigators hypothesize that each BCG vaccination will eliminate more and more of the disease causing white blood cells that could offer relief to the pancreas for increased survival and restoration of insulin secretion from the pancreas.

An additional adaptive trial for COVID-19 is also being conducted on these randomized double blinded type 1 diabetic subjects receiving BCG or placebo injections.

An expanded study arm has been approved for repeat dosing of BCG in adult Type I diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes treated continuously with insulin from time of diagnosis
* Age 18-65
* HIV antibody negative
* Normal CBC
* HCG negative (females)
* Anti-GAD Positive (except for subjects with c-peptide <10pmol/L)
* Fasting or stimulated c-peptide between 5-200 pmol/L
* Participation in protocol #2001P001379, "Autoimmunity: In Vitro Pathogenesis and Early Detection"

Exclusion Criteria:

* History of chronic infectious disease such as HIV or hepatitis
* History of tuberculosis, TB risk factors, positive interferon-gamma release assay (IGRA, also known as the T-SPOT.TB test), or BCG vaccination
* Current treatment with glucocorticoids (other than intermittent nasal or eye steroids), or disease or condition likely to require steroid therapy
* Other conditions or treatments associated with increased risk of infections such as patients with a previous history of severe burns, or treatment with immunosuppressive medications of any type (e.g. imuran, methotrexate, cyclosporine, etanercept, infliximab) for any reason
* Current treatment with aspirin > 160 mg/day or chronic, daily NSAIDs
* Current treatment with antibiotics
* History of keloid formation
* Average HbA1c over the past 5 years (or since diagnosis if duration is less than 5 years) <6.5 or > 8.5%
* History or evidence of chronic kidney disease (serum creatinine > 1.5mg/dL)
* History of proliferative diabetic retinopathy that has not been treated with laser therapy
* History of neuropathy, foot ulcers, amputations, or kidney disease
* Pregnant or not using acceptable birth control
* Living with someone who is immunosuppressed and/or at high risk for infectious diseases (for example HIV+ or taking immunosuppressive medications for any reason)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-06; Primary Completion 2029-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c values in juvenile onset type 1 diabetics | 1, 2, 3, 4, and 5 years after initial BCG/placebo injection
  A change in the hemoglobin A1c (HbA1c) measurement compared to self

SECONDARY OUTCOMES:
Insulin use in juvenile onset type 1 diabetics (AOO<21 years) | 4 weeks and 1, 2, 3, 4, and 5 years after initial BCG/placebo injection
  A change in insulin (IDAA1c) use as reported at study visits compared to self in juvenile onset type 1 diabetes.
Endogenous insulin levels in the blood in juvenile onset type 1 diabetics (AOO<21 years) | 4 weeks and 1, 2, 3, 4, and 5 years after initial BCG/placebo injection
  A change in c-peptide and proinsulin levels (as an analog for endogenous insulin) in the blood compared to self.
Autoimmunity in juvenile onset type 1 diabetes (AOO<21 years) | 4 weeks and 1, 2, 3, 4, and 5 years after initial BCG/placebo injection
  A change in autoantibodies and autoreactive T cells to monitor the drug mechanism for autoimmune changes.

OTHER OUTCOMES:
Exploratory: A Change in the above primary and secondary endpoints with Latent Autoimmune diabetes of adults (LADA; [a.k.a. Type 1.5 diabetes]; AOO>21 years) | 4 weeks and 1, 2, 3, 4, and 5 years after initial BCG/placebo injection
  A change in values as compared to self for participants with AOO>21 years of age.
COVID-19 and BCG Adaptive Study: Number of Type 1 Diabetics with COVID-19 symptomatic infections | 15 months beginning January 2020
  Number of symptomatic COVID-19 infections determined through PCR and antibody testing and symptoms collected through surveys and visits.
COVID-19 and BCG Adaptive Study: Impact of COVID-19 (severity, duration of symptoms, absence from work) | 15 months beginning January 2020
  A different severity of symptoms, duration of symptoms or absence from work for COVID-19 positive patients in the BCG or Placebo group.
COVID-19 and BCG Adaptive Study: Reported Rates of Infectious Diseases | 15 months beginning January 2020
  Rate of reported infectious disease adverse events categorized through MedDRA codes between the BCG and Placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Denise L Faustman, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Immunobiology Labs CNY 149, Charlestown, Massachusetts, United States

REFERENCES:
- [Derived] Faustman DL, Lee A, Hostetter ER, Aristarkhova A, Ng NC, Shpilsky GF, Tran L, Wolfe G, Takahashi H, Dias HF, Braley J, Zheng H, Schoenfeld DA, Kuhtreiber WM. Multiple BCG vaccinations for the prevention of COVID-19 and other infectious diseases in type 1 diabetes. Cell Rep Med. 2022 Sep 20;3(9):100728. doi: 10.1016/j.xcrm.2022.100728. Epub 2022 Aug 15. PMID 36027906
- See also: Faustman Lab Research Website — http://faustmanlab.org/